CLINICAL TRIAL: NCT06271343
Title: Non-interventional Single-center Study of the Contribution of DP8α Regulatory T Cells Induced by a Gut Microbiota Bacterium to Kidney Transplant Tolerance.
Brief Title: Kidney Graft Tolerance KTOL
Acronym: KTOL
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC23_0394
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Kidney Transplant Tolerance
Keywords: DP8 Regulatory Lymphocytes; Intestinal Microbiota; Tolerance; Transplant; Kidney

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Donor patients
- Recipient patients

SUMMARY:
Prospective experimental study using PBMC from a limited number of adult patients (15) treated at Nantes University Hospital for a kidney transplant from a related living donor.

The study will be carried out on PBMC from both donors and recipients, collected during visits scheduled as part of the clinical management of the donor/recipient pair.

The study will test the hypothesis that DP8α Tregs expressing CD73, whose frequency in blood increases stably after non-rejected kidney transplants, but not when patients have undergone or will subsequently undergo rejection, are enriched in donor-specific cells, which would be a strong argument in favor of a direct role for these Tregs in preventing transplant rejection, through their ability to inhibit immune responses directed against donor alloantigens.

ELIGIBILITY:
Inclusion Criteria:

* Adult donor-recipient pair.
* First or second kidney transplant from a related ABO-compatible living donor.
* BMI < 35 for recipients.
* Adult patients.
* Patients weighing over 50 kgs.

Exclusion Criteria:

* Donor/recipient ABO incompatibility
* BMI > 35 for recipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will use PBMCs from 15 patients receiving a kidney transplant from a living, ABO-compatible donor from their family or acquaintance. These PBMC will be obtained from blood samples taken before and 3 months after transplantation, in the context of normal patient management. The study will also use PBMC from the donor, taken before the transplant.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
To test the role of donor-specific DP8α Tregs in preventing kidney transplant rejection. | 3 months
  Measurement at D0 and 3 months post-transplant, and comparison, of the frequency of DP8a Tregs expressing CD73 among circulating T lymphocytes and the frequency of donor-reactive DP8a Tregs (identified in culture by their proliferative response to donor monocytes and clonal validation of DP8a Treg anti-donor reactivity at the 3-month post-transplant stage.

SECONDARY OUTCOMES:
Determine whether the increased anti-donor reactivity of the patient's DP8α Tregs after transplantation results from the amplification among them of clones and establish, if possible, the anti-donor reactivity of amplified clones. | 3 months
  Sorting of DP8a Tregs from the patient's blood before transplantation (D0) and at 3 months post-transplant, comparison of the TCR repertoire (TRA and TRB) of Tregs between these two stages, by a service provider. Identification (if possible by their Vb) of donor-reactive clones among the amplified TCR clones.
Determine whether clones of DP8α Tregs (reactive or not to donor antigens) are reactive to F. prausnitzii bacteria. | 3 months
  The response (proliferation or cytokine secretion) of donor-reactive DP8α Tregs clones will be tested against patient monocytes loaded with F. prausnitzii bacteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France